CLINICAL TRIAL: NCT01294410
Title: A Phase IIb Randomized, Placebo-Controlled Study to Evaluate the Clinical Efficacy and Safety of Induction and Maintenance Therapy With BMS-936557 in Subjects With Active Ulcerative Colitis (UC)
Brief Title: Induction and Maintenance Study of BMS-936557 Patients With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM129-005; 2010-022506-41 (EudraCT Number)
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1: Induction (Experimental): Placebo or Anti-IP-10 Antibody
  Interventions: Drug: Placebo; Drug: Anti-IP-10 Antibody
- Cohort 2: Induction (Experimental): Placebo or Anti-IP-10 Antibody
  Interventions: Drug: Placebo; Drug: Anti-IP-10 Antibody
- Cohort 3: Induction (Experimental): Placebo or Anti-IP-10 Antibody
  Interventions: Drug: Placebo; Drug: Anti-IP-10 Antibody
- Maintenance (Experimental): Placebo or Anti-IP-10 Antibody
  Interventions: Drug: Placebo; Drug: Anti-IP-10 Antibody
- Open Label (Other)
  Interventions: Drug: Anti-IP-10 Antibody

INTERVENTIONS:
Drug: Placebo — Normal Saline, Intravenous, 0mg, Once a week for the first two weeks and every other week thereafter, 7 Weeks
  Arms: Cohort 1: Induction; Cohort 2: Induction; Cohort 3: Induction
Drug: Placebo — Normal Saline, Intravenous, 0 mg, Every other week, Up to 757 days
  Arms: Maintenance
Drug: Anti-IP-10 Antibody — Solution for IV administration, Intravenous, 15 mg/kg, Once a week for the first two weeks and every other week thereafter, 7 weeks
  Arms: Cohort 1: Induction; Cohort 3: Induction
Drug: Anti-IP-10 Antibody — Solution for IV administration, Intravenous, 25 mg/kg, Once a week for the first two weeks and every other week thereafter, 7 weeks
  Arms: Cohort 2: Induction; Cohort 3: Induction
Drug: Anti-IP-10 Antibody — Solution for IV administration, Intravenous, 5 mg/kg, Every other week, Up to 757 days
  Arms: Maintenance
Drug: Anti-IP-10 Antibody — Intravenous, Solution for IV administration, 10 mg/kg, Every other week, Up to 757 days
  Arms: Maintenance
Drug: Anti-IP-10 Antibody — Intravenous, Solution for IV administration, 20 mg/kg, Every other week, Up to 757 days
  Arms: Maintenance
Drug: Anti-IP-10 Antibody — Intravenous, Solution for IV administration, 15 mg/kg or optimal dose, Every other week. Open
  Arms: Open Label

SUMMARY:
The purpose of this study is to determine whether BMS-936557 is effective in the treatment of moderate to severely active ulcerative colitis in patients who have had insufficient response and/or intolerance to other medical therapy for ulcerative colitis

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe UC confirmed by endoscopic and histologic evidence
* Mayo score ≥6 with an endoscopic subscore of ≥2
* Inadequate response and/or intolerance to one or more conventional therapy (i.e. oral aminosalicylates, immunosuppressants, corticosteroids, and/or TNF antagonist)

Exclusion Criteria:

* Diagnosis of Crohn's Disease or Indeterminate Colitis
* Diagnosis of UC that is limited to the rectum
* Evidence of fulminant colitis, toxic megacolon, or bowel perforation
* Current need for a colostomy or ileostomy
* Previous total or subtotal colectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Proportion of the subjects with clinical remission (defined as Mayo score ≤ 2 points with no individual subscore > 1 point) of BMS-936557 with that of the placebo | End of Induction [Week 11, Induction Period-78 (IP-78)]

SECONDARY OUTCOMES:
Proportion of the subjects with clinical response of BMS-936557 with that of the placebo | IP-78 (Week 11)
  Defined as a reduction from baseline in Mayo score ≥3 points and ≥30% and decrease from baseline in rectal bleeding subscore ≥1 point or absolute rectal bleeding subscore ≤1 point
Proportion of subjects with mucosal healing (defined as endoscopy subscore of ≤1 point) of BMS-936557 with that of the placebo | IP-78 (Week 11)
Proportion of subjects reporting Adverse event (AE), Serious adverse events (SAEs), AEs leading to discontinuation, and markedly abnormal laboratory values | IP-78 (Week 11)
Mean change from baseline at Inflammatory Bowel Disease Questionnaire (IBDQ) of subjects treated with BMS-936557 and placebo | Baseline (IP-1, Week 1) and IP-78 (Week 11)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (70):
- United States (23):
  - University Of California, San Diego, La Jolla, California
  - Santa Monica Research Institute, Santa Monica, California
  - Western States Clinical Research Inc., Wheat Ridge, Colorado
  - University Of Florida, Gainesville, Florida
  - Shafran Gasteroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Health Science Research Center, Pratt, Kansas
  - University Of Kentucky, Lexington, Kentucky
  - University Of Louisville, Louisville, Kentucky
  - Gastroenterology Research Of New Orleans, Hammond, Louisiana
  - Metropolitan Gastroenterology Group, Pc, Chevy Chase Cr, Chevy Chase, Maryland
  - Minnesota Gastroenterology, Pa, Plymouth, Minnesota
  - Westglen Gastrointestinal Consultants, Lee's Summit, Missouri
  - Long Island Clinical Research Assoc., Llp, Great Neck, New York
  - Mount Sinai School Of Medicine, New York, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Charlotte Gastroenterology & Hepatology, Pllc, Charlotte, North Carolina
  - Consultants For Clinical Research, Cincinnati, Ohio
  - Gastroenterology Research Of Lima, Lima, Ohio
  - Pharma Resource, East Providence, Rhode Island
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Gastroenterology Research Of San Antonio, San Antonio, Texas
  - Gastroenterology Research Of Tyler (Gerty), Tyler, Texas
- Australia (6):
  - Local Institution, Garran, Australian Capital Territory
  - Local Institution, Concord, New South Wales
  - Local Institution, Herston, Queensland
  - Local Institution, Parkville, Victoria
  - Local Institution, South Brisbane, Victoria
  - Local Institution, Fremantle, Western Australia
- Austria (2):
  - Local Institution, Graz
  - Local Institution, Vienna
- Belgium (3):
  - Local Institution, Bonheiden
  - Local Institution, Edegem
  - Local Institution, Leuven
- Brazil (3):
  - Local Institution, Goiânia, Goiás
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Botucatu, São Paulo
- Canada (4):
  - Local Institution, Calgary, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Kingston, Ontario
  - Local Institution, Vaughan, Ontario
- France (5):
  - Local Institution, Clichy
  - Local Institution, Lille
  - Local Institution, Nice
  - Local Institution, Pessac
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (3):
  - Local Institution, Hamburg
  - Local Institution, Kiel
  - Local Institution, Münster
- Hungary (3):
  - Local Institution, Budapest
  - Local Institution, Debrecen
  - Local Institution, Szeged
- Italy (4):
  - Local Institution, Padua
  - Local Institution, Roma
  - Local Institution, San Donato Milanese (mi)
  - Local Institution, San Giovanni Rotondo (fg)
- Mexico (5):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Mexico, D. F., Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Veracruz, Veracruz
- Netherlands (2):
  - Local Institution, Amsterdam
  - Local Institution, Rotterdam
- Poland (3):
  - Local Institution, Rzeszów
  - Local Institution, Sosnowiec
  - Local Institution, Warsaw
- South Africa (4):
  - Local Institution, Overport, KwaZulu-Natal
  - Local Institution, Claremont, Western Cape
  - Local Institution, Panorama, Western Cape
  - Local Institution, Paarl

REFERENCES:
- [Derived] Sandborn WJ, Colombel JF, Ghosh S, Sands BE, Dryden G, Hebuterne X, Leong RW, Bressler B, Ullman T, Lakatos PL, Reinisch W, Xu LA, Luo A. Eldelumab [Anti-IP-10] Induction Therapy for Ulcerative Colitis: A Randomised, Placebo-Controlled, Phase 2b Study. J Crohns Colitis. 2016 Apr;10(4):418-28. doi: 10.1093/ecco-jcc/jjv224. Epub 2015 Dec 30. PMID 26721935
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx